CLINICAL TRIAL: NCT04792021
Title: Effect of N-acetylcysteine on Oxidative Stress And Occurrence of Complications in Patients With COVID 19 Infections
Brief Title: Effect of N-acetylcysteine on Oxidative Stress in COVID-19 Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Misr International University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Sherkawy, Principal Investigator at the Faculty of pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-acetylcysteine in COVID 19
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Corona Virus Disease 19 (Covid19); Corona Virus Infection; Severe Acute Respiratory Syndrome Coronavirus 2(SARS-CoV2)
Keywords: N-acetylcysteine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
  One arm is the intervention arm: those receiving N-acetylcysteine (NAC). One arm is the control group : those not receiving N-acetylcysteine (NAC).
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-acetylcysteine (NAC) (Active Comparator): Patients receiving N-acetylcysteine (NAC)
  Interventions: Drug: N-acetylcysteine
- Control (No Intervention): Patients not receiving N-acetylcysteine (NAC)

INTERVENTIONS:
Drug: N-acetylcysteine — Oral formulation: 600 mg sachets of N-acetylcysteine
  Other Names: Acetylcysteine
  Arms: N-acetylcysteine (NAC)

SUMMARY:
The purpose of the study is to assess the potential therapeutic effect of N-acetylcysteine "NAC" in COVID 19 patients.

DETAILED DESCRIPTION:
This is a phase 3 trial enrolling subjects with newly diagnosed Corona virus disease 2019 ( COVID-19) infection who are classified as moderate cases and require hospitalization. Patients meeting eligibility criteria will be randomized either to receive oral N-acetylcysteine or not along with the institution treatment protocol . Treatment efficacy will be assessed using certain endpoints as follows:

1. Markers of inflammation and oxidative stress
2. Length of hospital stay
3. Need for ventilation
4. Mortality rate

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged more than 18 years
2. Documented COVID-19 infection (either performed on site or documented external report), only moderate cases will be included

Exclusion Criteria:

1. Known allergy or hypersensitivity to NAC
2. Pregnancy
3. Critically ill or mechanically ventilated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in TNF alfa level from baseline | from enrollment till the end of treatment at 2 weeks or until hospital discharge or death
  The mean change in TNF alfa is used to assess NAC efficacy

SECONDARY OUTCOMES:
Change in IL-6 level from baseline | from enrollment till the end of treatment at 2 weeks or until hospital discharge or death
  The mean change in IL-6 level is used to assess NAC efficacy
Change in glutathione peroxidase level from baseline | from enrollment till the end of treatment at 2 weeks or until hospital discharge or death
  The mean change in glutathione peroxidase is used to assess NAC efficacy
Length of hospital stay | Through study completion ( average 9 months)
  Duration of hospital stay for admitted patients
Need for mechanical ventilation | Through study completion ( average 9 months)
  Whether a patient required mechanical ventilation (intubation) or not

CONTACTS AND LOCATIONS:
Overall Officials: Sara M. Sherkawy, B.S.P, Principal Investigator — Misr International University; Lamia El Wakeel, Professor, Study Chair — Ain Shams University; Mona Schaalan, Professor, Study Director — Misr International University; Ayman Moharram, Professor, Study Director — El Kasr El Einy Hospital
Locations (1):
- Al Assema Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided